CLINICAL TRIAL: NCT05966597
Title: Effectiveness of Written Behavioural Persuasion Technique Intervention for Hypertension Management Among The Untreated Hypertension Population of The Community Observatory in Segamat, Johor: a 2-arm Randomised Controlled Trial Within Cohort
Brief Title: Written Behavioural Persuasion Technique Intervention for Hypertension Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University Malaysia (Other)
Collaborators: Monash University (Other)
Responsible Party: Principal Investigator, Tin Tin Su, Director of SEACO & Professor Global Public Health, Monash University Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MUHREC38735
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Behavior and Behavior Mechanisms
MeSH Terms: conditions — Hypertension; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Written persuasive leaflet (Experimental): Participants will receive a written persuasive leaflet in addition to the standard referral leaflet.
  Interventions: Behavioral: Written persuasive leaflet; Behavioral: Standard referral leaflet
- Standard referral leaflet (Sham Comparator): Participants will receive a standard referral leaflet.
  Interventions: Behavioral: Standard referral leaflet

INTERVENTIONS:
Behavioral: Written persuasive leaflet — Additional written behavioural persuasive technique leaflet and a standard referral leaflet provided at the end of the home-based health screening.
  Arms: Written persuasive leaflet
Behavioral: Standard referral leaflet — Standard referral leaflet provided at the end of the home-based health screening.

SUMMARY:
This study aims to examine the feasibility and effectiveness of written behavioural persuasion techniques intervention to encourage treatment initiation and follow-up for hypertension management among the untreated hypertension population of the SEACO cohort.

DETAILED DESCRIPTION:
Each household is given a unique identifier called house_id in the SEACO database. The randomisation will be computer-generated according to their house_id with a ratio of 1:1. During the house visit, participants' blood pressure will be taken three times, and the final reading will be the average of the second and third readings. Participants will be assessed based on the inclusion and exclusion criteria, i.e., age 35 years and above, blood pressure reading and reported not being diagnosed with or treated for hypertension. At the end of the house visit, all participants will receive a standard referral leaflet, and participants randomised to the intervention group will receive an additional written behavioural persuasion leaflet.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 and above
* Systolic blood pressure equal to or more than 140 mmHg
* Diastolic blood pressure equal to or more than 90 mmHg
* reported not being diagnosed with hypertension OR not being treated for hypertension

Exclusion Criteria:

* Involve in other research projects
* decline to participate/reject

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 893 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who see a doctor because of high blood pressure | Follow-up after 4-6 weeks receiving the leaflet
  The number of participants who see a doctor because of high blood pressure
Participants' intention to go see the doctor about their blood pressure (6-point Likert scale) | Follow-up after 4-6 weeks receiving the leaflet
  6-point Likert scale (strongly agree, moderately agree, somewhat agree, somewhat disagree, moderately disagree, strongly disagree) to measure participants' intention to go see the doctor about their blood pressure - "I intend to go to the doctor about my blood pressure", "I plan to go to the doctor about my blood pressure", "I want to go to the doctor about my blood pressure")
Participants' awareness of receiving the written communication during the health visit and their perceptions of the leaflets (6-point Likert scale) | Follow-up after 4-6 weeks receiving the leaflet
  6-point Likert scale (strongly agree, moderately agree, somewhat agree, somewhat disagree, moderately disagree, strongly disagree) to measure participants' awareness of receiving the leaflets during the health visit and their perceptions of the leaflets' content, usefulness, impact on seeking medical attention, and aesthetic appeal - "The leaflets contain useful information", "The leaflet was helpful. It made it easier for me to see a doctor and manage my blood pressure/ It would make it easier for me to see a doctor and manage my blood pressure", "The leaflet was persuasive. It made me want to see a doctor for my blood pressure", "I like the colour and design of the leaflet".
12-item Health Literacy score | Follow-up after 4-6 weeks receiving the leaflet
  12-item Health Literacy is a validated, self-reported instrument used to measure health literacy (HL). The index value for HL is obtained where 0 represents the lowest HL and 50 the highest HL

SECONDARY OUTCOMES:
Time taken for clinic visit (week) | Follow-up after 4-6 weeks receiving the leaflet
  Time taken (week) for participants to go see a doctor because of high blood pressure after receiving the leaflet
Blood pressure status during clinic visit | Follow-up after 4-6 weeks receiving the leaflet
  Participants' self-reported blood pressure status during the visit to the clinic/doctor (low, normal, high)

CONTACTS AND LOCATIONS:
Overall Officials: Tin Tin Su, Principal Investigator — Monash University Malaysia
Locations (1):
- South East Asia Community Observatory, Monash University Malaysia, Segamat, Johor, Malaysia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available. The MUHREC requirement to comply with the term "Retention and storage of data - The Chief Investigator is responsible for the storage and retention of the original data pertaining to the project for a minimum period of five years".

REFERENCES:
- [Background] Duong TV, Aringazina A, Kayupova G, Nurjanah, Pham TV, Pham KM, Truong TQ, Nguyen KT, Oo WM, Su TT, Majid HA, Sorensen K, Lin IF, Chang Y, Yang SH, Chang PWS. Development and Validation of a New Short-Form Health Literacy Instrument (HLS-SF12) for the General Public in Six Asian Countries. Health Lit Res Pract. 2019 Apr 10;3(2):e91-e102. doi: 10.3928/24748307-20190225-01. eCollection 2019 Apr. PMID 31294310